CLINICAL TRIAL: NCT00004152
Title: A Pilot Study to Compare 18F-Fluorodeoxyglucose Positron Emission Tomography (PET) Scanning in Addition to CT Scanning With CT Scanning Alone in the Pre-Operative Evaluation of Patients With Stage III and IV Melanoma
Brief Title: PET and CT Scans to Evaluate Patients With Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: 99-004; MSKCC-99004; NCI-G99-1619
Record Dates: First submitted 1999-12-10; First posted 2004-02-16 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18

INTERVENTIONS:
Drug: iodinated contrast dye
Procedure: computed tomography
Procedure: positron emission tomography
Radiation: fludeoxyglucose F 18

SUMMARY:
RATIONALE: Diagnostic procedures may improve the ability to detect metastatic melanoma and to determine the extent of disease.

PURPOSE: Phase II trial to evaluate the effectiveness of PET and CT scans to detect metastatic disease in patients who have stage III or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the sensitivity, specificity, and accuracy of fludeoxyglucose F 18 (FDG) positron emission tomography (PET) imaging in detecting metastatic disease in patients with stage III or IV melanoma considered for operative management based on the currently accepted diagnostic work up including CT imaging. II. Determine how often the clinical management of these patients is altered based on FDG PET imaging findings in addition to CT scan results.

OUTLINE: Patients are required to fast for a minimum of 6 hours prior to positron emission tomography (PET) imaging. Fludeoxyglucose F 18 (FDG) is administered IV over 15 minutes followed 50-60 minutes later by whole body PET imaging. Iodinated contrast dye is administered by IV injection and by mouth followed by CT imaging of the chest, abdomen, and pelvis within 2 weeks of PET imaging. Whole body FDG PET imaging and CT imaging of the chest, abdomen, and pelvis are repeated at 6 months. Initial positive PET or CT imaging results are verified based on surgical and/or biopsy findings or clinical follow-up.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven melanoma considered for operative management with 1 of the following: Deep primary melanoma (greater than 4 mm, stage IIIA) Regional nodal disease (stage IIIB) Locally or regionally recurrent disease of an extremity considered for operative resection or isolated limb perfusion with curative intent Systemic disease considered for curative resection (stage IV)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Not pregnant or nursing Fertile patients must use effective contraception Able to fast for 6 hours Able to lie still for positron emission tomography imaging No second malignancy except previously treated nonmelanomatous skin cancer or carcinoma in situ of the cervix No active infection No inflammatory disease (sarcoidosis or rheumatoid arthritis) No allergy to shellfish or contrast dye used for CT imaging

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-02; Primary Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary S. Brady, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States